CLINICAL TRIAL: NCT02634684
Title: Pharmacologic Augmentation of Neurocognition and Cognitive Training in Psychosis
Brief Title: Pharmacologically-augmented Cognitive Therapies (PACTs) for Schizophrenia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Neal R. Swerdlow, M.D., Ph.D., Professor of Psychiatry and Director of the Research Residency Track at the University of California, San Diego, School of Medicine., University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5R01MH059803-15 (NIH); Eyeblink Study (Other: UC San Diego)
Record Dates: First submitted 2015-12-14; First posted 2015-12-18 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizoaffective Disorder; Mental Disorders; Anti-Dyskinesia Agents; Antiparkinson Agents; Central Nervous System Agents; Dopamine Agents; Excitatory Amino Acid Agents; Excitatory Amino Acid Antagonists; Molecular Mechanisms of Pharmacological Action; Neurotransmitter Agents; Pharmacologic Actions; Physiological Effects of Drugs; Therapeutic Uses; Prepulse inhibition; Neurocognition; Working memory; Dextroamphetamine; MATRICS Consensus Cognitive Battery; Pharmacologic Augmentation of Cognitive Therapies; Sensory discrimination learning; Targeted Cognitive Training; rs4680 polymorphism of catechol-O-methyltransferase (COMT)
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dextroamphetamine (Active Comparator): Drug: Dexedrine, dextroamphetamine, d-amphetamine.
  Dosage form, frequency and duration: Each participant receives a single pill of placebo or active drug (dextroamphetamine 10 mg) 30 minutes after arriving at the lab. The participant then completes approximately 6 hours of testing in the laboratory. The participant stays at the lab for 7.5 hours in order to monitor physical condition in case the participant received the active pill One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.
  Interventions: Drug: Dextroamphetamine; Drug: Placebo
- Placebo (Placebo Comparator): Drug: Dexedrine, dextroamphetamine, d-amphetamine
  Dosage form, frequency and duration: Each participant receives a single pill of placebo or active drug (dextroamphetamine 10 mg) 30 minutes after arriving at the lab. The participant then completes approximately 6 hours of testing in the laboratory. The participant stays at the lab for 7.5 hours in order to monitor physical condition in case the participant received the active pill One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.
  Interventions: Drug: Dextroamphetamine; Drug: Placebo

INTERVENTIONS:
Drug: Dextroamphetamine — Each participant receives a single pill of placebo or active drug (dextroamphetamine 10 mg) and completes approximately 6 hours of testing in the laboratory. One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.
  Other Names: d-amphetamine; Dexedrine
Drug: Placebo — Each participant receives a single pill of placebo or active drug (dextroamphetamine 10 mg) and completes approximately 6 hours of testing in the laboratory. One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.

SUMMARY:
This application seeks renewed support for MH59803, "Dopaminergic substrates of startle gating across species," to extend a clear path of "bench-to-bedside" progress towards a critical paradigm shift in therapeutic models for schizophrenia (SZ) and schizoaffective disorder, depressed type (SZA): the use of Pharmacologic Augmentation of Cognitive Therapies (PACTs). This novel therapeutic strategy for SZ/SZA directly addresses the need for more effective treatments for this devastating disorder. MH59803 has investigated the neural regulation of laboratory-based measures of deficient information processing in SZ/SZA patients, using rodents and healthy human subjects (HS) to explicate the biology of these deficits, and to establish a rational basis for developing novel therapies for SZ/SZA. In its first 9 years, MH59803 studies of the neural regulation of prepulse inhibition (PPI) of startle in rats focused on basic neurobiological and molecular mechanisms. Over the past 2 years of support, MH59803 studies moved "from bench-to-bedside," focusing on dopamine (DA) agonist effects on PPI and neurocognition in HS, and their regulation by genes identified in cross-species studies. These studies detected biological markers that predict PPI-enhancing and pro-cognitive effects of the DA releaser, amphetamine (AMPH) in humans, leading to specific predictions of AMPH effects on PPI, neurocognition and Targeted Cognitive Training in SZ/SZA patients. If confirmed in the present application, these predictions could help transform therapeutic approaches to SZ/SZA. This renewal application of MH59803 thus reflects a logical progression of studies at systems and molecular levels, translated first to HS, and now to potentially transformative therapeutic models in SZ/SZA patients.

DETAILED DESCRIPTION:
MH59803 demonstrated that AMPH (20 mg p.o.) significantly increased PPI and neurocognitive performance (MATRICS Consensus Cognitive Battery; MCCB) in HS characterized by specific performance-based or genetic biomarkers, including the val/val genotype for the rs4680 polymorphism of catechol-O-methyltransferase (COMT). Mechanistically-informative results were detected in studies of AMPH effects on PPI in rats with high vs. low brain regional Comt expression. Together with several reports of improved neurocognition and no adverse effects of acute or sustained AMPH administration to antipsychotic (AP)-medicated SZ/SZA patients, MH59803 findings provide a strong rationale for the next goal of this application: to test the potential utility of AMPH in a paradigm of biomarker-informed "PACTs". This "next step" is highly innovative - never previously reported, or perhaps even attempted - and consistent with National Institute of Mental Health (NIMH) objectives, directly challenges existing models for SZ/SZA therapeutics. Investigators will determine whether a test dose of 10 mg AMPH p.o. administered to biomarker-identified, AP-medicated SZ/SZA patients generates predicted increases in PPI, MCCB performance, and sensory discrimination learning in a Targeted Cognitive Training (TCT) module. In total, Investigators will leverage knowledge generated through converging cross-species studies in MH59803, to directly advance scientific and clinical domains, by testing the effects of a pro-cognitive drug on neurophysiological and neurocognitive performance, and Targeted Cognitive Training, in biomarker-stratified subgroups of SZ/SZA patients.

Aim: To assess acute effects of AMPH (0 vs 10 mg po) on PPI, neurocognition and computerized TCT in AP-medicated SZ/SZA patients. Hypothesis: PPI- and MCCB-enhancing effects of AMPH seen previously in HS will also be detected in SZ/SZA patients, as will TCT-enhancing effects of AMPH. Prediction: In a within-subject, placebo-controlled, randomized design, AMPH (10 mg po) will increase PPI and enhance MCCB and TCT performance in medicated SZ/SZA patients, particularly among those characterized by low basal performance levels and/or the val/val rs4680 COMT polymorphism. Concurrent HS testing will confirm and extend findings of AMPH effects on PPI and neurocognition, and help interpret findings in SZ/SZA patients.

In all participants, the aim to assess acute effects of 0 vs. 10 mg po dextroamphetamine (AMPH) on Prepulse Inhibition (PPI), neurocognition MATRICS: Consensus Cognitive Battery; MCCB, and computerized Targeted Cognitive Training (TCT).

Hypothesis: AMPH will enhance:

1. PPI
2. neurocognition (MCCB performance)
3. computerized TCT performance in biomarker-identified SZ/SZA patients.
4. The PPI and MCCB-enhancing effects of AMPH seen previously in HS will also be detected in SZ/SZA patients, as will TCT-enhancing effects of AMPH.

Prediction: In a within-subject, placebo-controlled, randomized design, AMPH (10 mg po) will increase PPI and enhance MCCB and TCT performance in medicated SZ/SZA patients, particularly among those characterized by low basal performance levels and/or the val/val rs4680 COMT polymorphism. Concurrent HS testing will confirm and extend findings of AMPH effects on PPI and neurocognition, and help interpret findings in SZ/SZA patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old:
* Drug Free (No recreational/street drugs)
* Diagnosis of Schizophrenia or Schizoaffective Disorder, Depressed Type
* Must be stable on antipsychotic medication for at least 1 month
* Any medications other than antipsychotic medications need to be stable for at least 1 week

Exclusion Criteria:

* Dominant hand injury
* Hearing impairment at 40 dB
* Irregular menstrual cycle or cycle is no within in 25-35 days (menopausal is eligible)
* EKG, conduction abnormalities confirmed by cardiologist
* Reading component of Wide Range Achievement Test 4 (WRAT4) Score less than 70
* Any serious illness, including: Insulin-dependent diabetes, HIV, AIDS, cancer, stroke, heart attack, uncontrolled hypothyroidism
* Sleep apnea
* A diagnosis of epilepsy or history of seizures with loss of consciousness
* Open/closed head injury with loss of consciousness greater than 1 minute at any time in the lifetime
* Blood pressure: Systolic Blood Pressure < 90 or > 160, Diastolic Blood Pressure < 45 or > 95
* Heart Rate < 55 or > 110
* Current use of Dexatrim or drugs containing phenylephrine (eligible if not used for at least 72 hours prior to participation)
* Current use of St. John's Wort, Milk Thistle (eligible if for at least 1 month)
* Self report of any illicit drug use within the last 30 days
* Positive urine toxicology
* Self-report of any use of ecstasy, lysergic acid diethylamide (LSD), mushrooms, gamma hydroxybutyrate (GHB), ketamine, phencyclidine (PCP), heroin or any intravenous-drugs within past year
* If there is a history of substance abuse/addiction, participant must be in remission for at least 6 months
* Within 1 month of recent psychiatric hospitalization
* Current mania
* Dementia/Alzheimer's diagnosis
* Mania episode meeting criteria outlined in the MINI-International Neuropsychiatric Interview Plus 6.0 (M.I.N.I. plus 6.0) anytime in the lifetime (hypomania/Bipolar II eligible)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal R. Swerdlow, M.D., Ph.D., Principal Investigator — UC San Diego
Locations (1):
- Clinical Teaching Facility (CTF-B102) at UCSD Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swerdlow NR. Beyond antipsychotics: pharmacologically-augmented cognitive therapies (PACTs) for schizophrenia. Neuropsychopharmacology. 2012 Jan;37(1):310-1. doi: 10.1038/npp.2011.195. No abstract available. PMID 22157876
- [Background] Barch DM, Carter CS. Amphetamine improves cognitive function in medicated individuals with schizophrenia and in healthy volunteers. Schizophr Res. 2005 Sep 1;77(1):43-58. doi: 10.1016/j.schres.2004.12.019. PMID 16005384
- [Background] Fisher M, Holland C, Merzenich MM, Vinogradov S. Using neuroplasticity-based auditory training to improve verbal memory in schizophrenia. Am J Psychiatry. 2009 Jul;166(7):805-11. doi: 10.1176/appi.ajp.2009.08050757. Epub 2009 May 15. PMID 19448187
- [Background] Fisher M, Holland C, Subramaniam K, Vinogradov S. Neuroplasticity-based cognitive training in schizophrenia: an interim report on the effects 6 months later. Schizophr Bull. 2010 Jul;36(4):869-79. doi: 10.1093/schbul/sbn170. Epub 2009 Mar 5. PMID 19269924
- [Background] Tarasenko M, Perez VB, Pianka ST, Vinogradov S, Braff DL, Swerdlow NR, Light GA. Measuring the capacity for auditory system plasticity: An examination of performance gains during initial exposure to auditory-targeted cognitive training in schizophrenia. Schizophr Res. 2016 Apr;172(1-3):123-30. doi: 10.1016/j.schres.2016.01.019. Epub 2016 Feb 2. PMID 26851143
- [Background] Vinogradov S, Fisher M, de Villers-Sidani E. Cognitive training for impaired neural systems in neuropsychiatric illness. Neuropsychopharmacology. 2012 Jan;37(1):43-76. doi: 10.1038/npp.2011.251. Epub 2011 Nov 2. PMID 22048465
- [Background] Chew ML, Mulsant BH, Pollock BG, Lehman ME, Greenspan A, Mahmoud RA, Kirshner MA, Sorisio DA, Bies RR, Gharabawi G. Anticholinergic activity of 107 medications commonly used by older adults. J Am Geriatr Soc. 2008 Jul;56(7):1333-41. doi: 10.1111/j.1532-5415.2008.01737.x. Epub 2008 May 26. PMID 18510583
- [Background] Chou HH, Talledo JA, Lamb SN, Thompson WK, Swerdlow NR. Amphetamine effects on MATRICS Consensus Cognitive Battery performance in healthy adults. Psychopharmacology (Berl). 2013 May;227(1):165-76. doi: 10.1007/s00213-012-2948-x. Epub 2013 Jan 12. PMID 23314393
- [Background] Lieberman JA, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Keefe RS, Davis SM, Davis CE, Lebowitz BD, Severe J, Hsiao JK; Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) Investigators. Effectiveness of antipsychotic drugs in patients with chronic schizophrenia. N Engl J Med. 2005 Sep 22;353(12):1209-23. doi: 10.1056/NEJMoa051688. Epub 2005 Sep 19. PMID 16172203
- [Background] Dinse HR, Ragert P, Pleger B, Schwenkreis P, Tegenthoff M. Pharmacological modulation of perceptual learning and associated cortical reorganization. Science. 2003 Jul 4;301(5629):91-4. doi: 10.1126/science.1085423. PMID 12843392
- [Background] Goldberg TE, Bigelow LB, Weinberger DR, Daniel DG, Kleinman JE. Cognitive and behavioral effects of the coadministration of dextroamphetamine and haloperidol in schizophrenia. Am J Psychiatry. 1991 Jan;148(1):78-84. doi: 10.1176/ajp.148.1.78. PMID 1984711
- [Background] Green MF. What are the functional consequences of neurocognitive deficits in schizophrenia? Am J Psychiatry. 1996 Mar;153(3):321-30. doi: 10.1176/ajp.153.3.321. PMID 8610818
- [Background] Green MF, Kern RS, Heaton RK. Longitudinal studies of cognition and functional outcome in schizophrenia: implications for MATRICS. Schizophr Res. 2004 Dec 15;72(1):41-51. doi: 10.1016/j.schres.2004.09.009. PMID 15531406
- [Background] Hamidovic A, Dlugos A, Palmer AA, de Wit H. Catechol-O-methyltransferase val158met genotype modulates sustained attention in both the drug-free state and in response to amphetamine. Psychiatr Genet. 2010 Jun;20(3):85-92. doi: 10.1097/YPG.0b013e32833a1f3c. PMID 20414144
- [Background] Hamidovic A, Dlugos A, Palmer AA, de Wit H. Polymorphisms in dopamine transporter (SLC6A3) are associated with stimulant effects of D-amphetamine: an exploratory pharmacogenetic study using healthy volunteers. Behav Genet. 2010 Mar;40(2):255-61. doi: 10.1007/s10519-009-9331-7. Epub 2010 Jan 21. PMID 20091113
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Keefe RS, Bilder RM, Davis SM, Harvey PD, Palmer BW, Gold JM, Meltzer HY, Green MF, Capuano G, Stroup TS, McEvoy JP, Swartz MS, Rosenheck RA, Perkins DO, Davis CE, Hsiao JK, Lieberman JA; CATIE Investigators; Neurocognitive Working Group. Neurocognitive effects of antipsychotic medications in patients with chronic schizophrenia in the CATIE Trial. Arch Gen Psychiatry. 2007 Jun;64(6):633-47. doi: 10.1001/archpsyc.64.6.633. PMID 17548746
- [Background] Kumari V, Premkumar P, Fannon D, Aasen I, Raghuvanshi S, Anilkumar AP, Antonova E, Peters ER, Kuipers E. Sensorimotor gating and clinical outcome following cognitive behaviour therapy for psychosis. Schizophr Res. 2012 Feb;134(2-3):232-8. doi: 10.1016/j.schres.2011.11.020. Epub 2011 Dec 3. PMID 22138048
- [Background] Mattay VS, Goldberg TE, Fera F, Hariri AR, Tessitore A, Egan MF, Kolachana B, Callicott JH, Weinberger DR. Catechol O-methyltransferase val158-met genotype and individual variation in the brain response to amphetamine. Proc Natl Acad Sci U S A. 2003 May 13;100(10):6186-91. doi: 10.1073/pnas.0931309100. Epub 2003 Apr 25. PMID 12716966
- [Background] Light GA, Swerdlow NR. Neurophysiological biomarkers informing the clinical neuroscience of schizophrenia: mismatch negativity and prepulse inhibition of startle. Curr Top Behav Neurosci. 2014;21:293-314. doi: 10.1007/7854_2014_316. PMID 24850080
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Pietrzak RH, Snyder PJ, Maruff P. Amphetamine-related improvement in executive function in patients with chronic schizophrenia is modulated by practice effects. Schizophr Res. 2010 Dec;124(1-3):176-82. doi: 10.1016/j.schres.2010.09.012. Epub 2010 Oct 13. PMID 20947305
- [Background] Pietrzak RH, Snyder PJ, Maruff P. Use of an acute challenge with d-amphetamine to model cognitive improvement in chronic schizophrenia. Hum Psychopharmacol. 2010 Jun-Jul;25(4):353-8. doi: 10.1002/hup.1118. PMID 20521327
- [Background] Ressler KJ, Rothbaum BO, Tannenbaum L, Anderson P, Graap K, Zimand E, Hodges L, Davis M. Cognitive enhancers as adjuncts to psychotherapy: use of D-cycloserine in phobic individuals to facilitate extinction of fear. Arch Gen Psychiatry. 2004 Nov;61(11):1136-44. doi: 10.1001/archpsyc.61.11.1136. PMID 15520361
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Shilling PD, Saint Marie RL, Shoemaker JM, Swerdlow NR. Strain differences in the gating-disruptive effects of apomorphine: relationship to gene expression in nucleus accumbens signaling pathways. Biol Psychiatry. 2008 Apr 15;63(8):748-58. doi: 10.1016/j.biopsych.2007.10.015. Epub 2008 Feb 20. PMID 18083141
- [Background] Swerdlow NR. Are we studying and treating schizophrenia correctly? Schizophr Res. 2011 Aug;130(1-3):1-10. doi: 10.1016/j.schres.2011.05.004. Epub 2011 Jun 8. PMID 21645998
- [Background] Swerdlow NR, Bhakta S, Chou HH, Talledo JA, Balvaneda B, Light GA. Memantine Effects On Sensorimotor Gating and Mismatch Negativity in Patients with Chronic Psychosis. Neuropsychopharmacology. 2016 Jan;41(2):419-30. doi: 10.1038/npp.2015.162. Epub 2015 Jun 11. PMID 26062785
- [Background] Swerdlow NR, Light GA, Sprock J, Calkins ME, Green MF, Greenwood TA, Gur RE, Gur RC, Lazzeroni LC, Nuechterlein KH, Radant AD, Ray A, Seidman LJ, Siever LJ, Silverman JM, Stone WS, Sugar CA, Tsuang DW, Tsuang MT, Turetsky BI, Braff DL. Deficient prepulse inhibition in schizophrenia detected by the multi-site COGS. Schizophr Res. 2014 Feb;152(2-3):503-12. doi: 10.1016/j.schres.2013.12.004. Epub 2014 Jan 7. PMID 24405980
- [Background] Talledo JA, Sutherland Owens AN, Schortinghuis T, Swerdlow NR. Amphetamine effects on startle gating in normal women and female rats. Psychopharmacology (Berl). 2009 May;204(1):165-75. doi: 10.1007/s00213-008-1446-7. Epub 2009 Jan 16. PMID 19148623
- [Background] Turetsky BI, Calkins ME, Light GA, Olincy A, Radant AD, Swerdlow NR. Neurophysiological endophenotypes of schizophrenia: the viability of selected candidate measures. Schizophr Bull. 2007 Jan;33(1):69-94. doi: 10.1093/schbul/sbl060. Epub 2006 Nov 29. PMID 17135482
- [Background] Wilkinson GS, Robertson GJ (2006) WRAT4: Wide Range Achievement Test professional manual, 4th edn Psychological Assessment Resources: Lutz, FL

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Schizophrenia: Placebo 1st, Then 10 mg Amphetamine; Subjects With Schizophrenia: 10 mg Amphetamine 1st, Then Placebo; Healthy Subjects: Placebo 1st, Then 10 mg Amphetamine; Healthy Subjects: 10 mg Amphetamine 1st, Then Placebo: Drug: Dexedrine, dextroamphetamine, d-amphetamine.
  Dosage form, frequency and duration: Each participant receives a single pill of placebo or active drug (dextroamphetamine) 30 minutes after arriving at the lab. The participant then completes ~6 hours of testing in the laboratory. The participant stays at the lab for ~7.5 hours to monitor physical condition in case the participant received the active pill. One week later, the participant receives a single pill of comparator and is again tested in the laboratory. Total of 1 visits, approximately 1 week apart; in total, each participant receives one placebo pill and 1 active pill separated by one week.
  Dextroamphetamine: Each participant receives a single pill of placebo or active drug (dextroamphetamine 10 mg) and completes approximately 6 hours of testing in the laboratory. One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.
  Placebo: Each participant receives a single pill of placebo or active drug (dextroamphetamine 10 mg) and completes approximately 6 hours of testing in the laboratory. One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.
Period: Overall Study
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 10 mg Amphetamine | Subjects With Schizophrenia: 10 mg Amphetamine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 10 mg Amphetamine | Healthy Subjects: 10 mg Amphetamine 1st, Then Placebo
Started | 19 | 19 | 21 | 23
Completed | 19 | 19 | 21 | 23
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 10 mg Amphetamine | Subjects With Schizophrenia: 10 mg Amphetamine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 10 mg Amphetamine | Healthy Subjects: 10 mg Amphetamine 1st, Then Placebo | Total
Number analyzed (Participants) | 19 | 19 | 21 | 23 | 82
Age, Continuous [Mean (Full Range); unit: years] | 39 [23 to 51] | 42 [27 to 55] | 29 [19 to 55] | 30 [20 to 53] | 35 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 6 | 6 | 29
  Male | 8 | 13 | 15 | 17 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 6 | 5 | 24
  Not Hispanic or Latino | 12 | 9 | 13 | 18 | 52
  Unknown or Not Reported | 2 | 2 | 2 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 2 | 4 | 12
  Asian | 0 | 2 | 5 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 8 | 3 | 3 | 1 | 15
  White | 5 | 7 | 7 | 12 | 31
  More than one race | 2 | 2 | 1 | 0 | 5
  Unknown or Not Reported | 1 | 1 | 3 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 21 | 23 | 82

OUTCOME MEASURES:

1. Primary Outcome: Prepulse Inhibition (PPI)
Description: PPI was assessed with 42 trials of 6 types: 118 dB 40 ms pulse alone (P) & the same P preceded 10, 20, 30, 60, or 120 ms by a prepulse (pp) 16 dB over background. Startle magnitude (SM), habituation, latency & latency facilitation were measured to interpret changes in PPI.
  %PPI = 100 x [(SM on P trials) - (SM on pp+P trials)] / SM on P trials. Example:
  SM on P trials = 80 units SM on pp+P trials = 30 units %PPI = 100 x (80-30)/80 = 100 x 50/80 = 62.5%
  Greater %PPI mean the reflex has been inhibited to a greater extent in the presence of a pp.
  %PPI can't exceed 100: when SM on pp+P trials = 0, then %PPI = 100 x (SM on P trials - 0)/SM on P trials = 100 x 1 = 100%.
  However, %PPI can theoretically be infinitely negative since SM on pp+P trials could be infinitely large ("prepulse facilitiation" (PPF)), i.e. SM is potentiated in the presence of a pp. PPF is "normal" at very short & very long pp intervals, but not within a species-specific physiological range of intervals.
Time Frame: two visits, 1 week apart, each visit lasting approximately 6 hours
Measure: Mean (Standard Deviation); unit: % inhibition of startle
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 10 mg Amphetamine | Subjects With Schizophrenia: 10 mg Amphetamine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 10 mg Amphetamine | Healthy Subjects: 10 mg Amphetamine 1st, Then Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 23
% inhibition of startle
  Placebo | 22.629 (62.657) | 41.162 (42.103) | 50.626 (25.850) | 50.626 (29.621)
  Amphetamine | 32.656 (57.669) | 39.545 (33.429) | 45.822 (31.777) | 53.029 (24.671)

2. Secondary Outcome: MATRICS Consensus Cognitive Battery Performance (MCCB)
Description: The T-score indicates the performance on a neurocognitive battery of tests. Higher score reflects better performance.
Time Frame: two visits, 1 week apart, each visit lasting approximately 6 hours
Measure: Mean (Standard Deviation); unit: standardized T-score
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 10 mg Amphetamine | Subjects With Schizophrenia: 10 mg Amphetamine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 10 mg Amphetamine | Healthy Subjects: 10 mg Amphetamine 1st, Then Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 23
standardized T-score
  placebo | 31.895 (15.937) | 39.895 (11.704) | 54.476 (11.557) | 57.870 (11.153)
  amphetamine | 33.842 (16.269) | 38.105 (12.552) | 55.476 (11.383) | 56.000 (11.286)

3. Secondary Outcome: Targeted Cognitive Training (TCT): PositScience, Inc.
Description: Auditory discrimination learning: Subjects identify direction (up vs. down) of 2 consecutive sound sweeps. Parameters (e.g. inter-sweep interval, sweep duration) are established for subjects to maintain 80% correct responses. On screen and test days, subjects complete 1h of TCT. Analytic software yields the key measures: auditory processing speed (APS) and APS "learning". APS is the shortest inter-stimulus interval at which a subject performs to criteria and APS learning is the difference (ms) between the first APS and the best APS of the subsequent trials. A smaller APS reflects "better" discrimination (i.e., subject correctly identified frequency "sweep" direction despite a smaller ms gap between stimuli) and a larger ms value for APS learning reflects more learning, i.e., faster APS with repeated trials. Limits for APS are capped at 0-to-1000 ms; values for APS learning are capped at (-) 1000-to-APS.
Time Frame: two visits, 1 week apart, each visit lasting approximately 6 hours
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Subjects With Schizophrenia: Placebo 1st, Then 10 mg Amphetamine | Subjects With Schizophrenia: 10 mg Amphetamine 1st, Then Placebo | Healthy Subjects: Placebo 1st, Then 10 mg Amphetamine | Healthy Subjects: 10 mg Amphetamine 1st, Then Placebo
Number analyzed (Participants) | 19 | 19 | 21 | 23
msec
  placebo | -15.118 (346.088) | -50.158 (218.464) | 5.911 (75.105) | -2.113 (107.563)
  amphetamine | 52.647 (305.887) | 101.000 (434.379) | 35.905 (64.539) | 29.190 (83.183)

ADVERSE EVENTS:
Time Frame: two visits, 1 week apart, each visit lasting approximately 6 hours
Description: Each subject received both interventions (placebo (PBO) and 10 mg amphetamine (AMPH)) separated by 1 week (wk), with pill order (PBO wk 1, AMPH wk 2 vs. AMPH wk 1, PBO wk 2) balanced. The 2 groups were "Subjects with schizophrenia" (SZ) and "healthy subjects"(HS). Assuming that adverse effects are independent of test order, there are 4 possible Arms/Groups; adverse events across these 4 Arms/Groups were:
  SZ: AMPH = 0 SZ: PBO = 0 HS: AMPH = 0 HS: PBO = 0
Groups:
- Subjects With Schizophrenia: Placebo; Healthy Subjects: Placebo: Placebo: Each participant receives a single pill of placebo or active drug (dextroamphetamine 10 mg) and completes approximately 6 hours of testing in the laboratory. One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.
- Subjects With Schizophrenia: 10 mg Amphetamine; Healthy Subjects: 10 mg Amphetamine: Dextroamphetamine: Each participant receives a single pill of placebo or active drug (dextroamphetamine 10 mg) and completes approximately 6 hours of testing in the laboratory. One week later, that participant receives a single pill of the alternate comparator and is again tested in the laboratory. Thus, in total, each participant receives one placebo pill and one active pill, separated by one week.
Arm/Group | Subjects With Schizophrenia: Placebo | Subjects With Schizophrenia: 10 mg Amphetamine | Healthy Subjects: Placebo | Healthy Subjects: 10 mg Amphetamine
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT02634684/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT02634684/SAP_001.pdf